CLINICAL TRIAL: NCT02318810
Title: The Influence of the Neuromuscular Blockade on Mask Ventilation; a Placebo Controlled, Randomized Trial With Three Different Dosages of Rocuronium (0.3 mg/kg, 0.6 mg/kg and 0.9 mg/kg)
Brief Title: Influence of the Neuromuscular Blockade on Mask Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Thomas Mencke, Prof. Dr. Thomas Mencke, University of Rostock
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A 2014 1212
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Complication of Ventilation Therapy; Observation of Neuromuscular Block
Keywords: Muscle relaxants
MeSH Terms: conditions — Muscle Hypotonia | interventions — Rocuronium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Rocuronium 0.3 mg/kg (Active Comparator): Patients receive rocuronium 0.3 mg/kg
  Interventions: Drug: Rocuronium 0.3 mg/kg
- Rocuronium 0.6 mg/kg (Active Comparator): Patients receive rocuronium 0.6 mg/kg
  Interventions: Drug: Rocuronium 0.6 mg/kg
- Rocuronium 0.9 mg/kg (Active Comparator): Patients receive rocuronium 0.9 mg/kg
  Interventions: Drug: Rocuronium 0.9 mg/kg
- Placebo (Placebo Comparator): Patients receive saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rocuronium 0.3 mg/kg — Patients receive rocuronium 0.3 mg/kg
  Other Names: Esmeron
  Arms: Rocuronium 0.3 mg/kg
Drug: Rocuronium 0.6 mg/kg — Patients receive rocuronium 0.6 mg/kg
  Other Names: Esmeron
  Arms: Rocuronium 0.6 mg/kg
Drug: Rocuronium 0.9 mg/kg — Patients receive rocuronium 0.9 mg/kg
  Other Names: Esmeron
  Arms: Rocuronium 0.9 mg/kg
Drug: Placebo — Patients receive saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Mask ventilation during induction of anesthesia can be improved by administration of neuromuscular blocking agents (NMBAs). NMBAs are usually administered after testing mask ventilation; however, muscle relaxants may improve mask ventilation and they do not alter mask ventilation. Thus, growing evidence suggests to administer muscle relaxants before testing mask ventilation. We will study different dosages of rocuronium; we assume that higher dosages of rocuronium will improve mask ventilation compared with lower dosages.

DETAILED DESCRIPTION:
Mask ventilation during induction of anesthesia can be improved by administration of neuromuscular blocking agents (NMBAs). NMBAs are usually administered after testing mask ventilation; however, muscle relaxants may improve mask ventilation and they do not alter mask ventilation. Thus, growing evidence suggests to administer muscle relaxants before testing mask ventilation.We will administer rocuronium 0.3 mg/kg, 0.6 mg/kg, 0.9 mg/kg and saline (placebo group) before starting with mask ventilation. We will grade mask ventilation based on various scores before and after rocuronium application. Afterwards patient's tracheas will be intubated. We assess risk factors for difficult mask ventilation.

We hypothesize that rocuronium 0.9 mg/kg will be superior to rocuronium 0.3 mg/kg and saline.

ELIGIBILITY:
Inclusion Criteria:

* patients with ASA I-III
* required tracheal intubation
* informed consent

Exclusion Criteria:

* known allergy against anesthetics
* known difficult airway

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of improved mask ventilation after rocuronium administration | Two minutes after rocuronium administration
  Graded with various scores

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mencke, Prof., Principal Investigator — University of Rostock
Locations (1):
- Department of Anesthesia and Intensive Care Medicine, University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: Undecided